CLINICAL TRIAL: NCT03144219
Title: A Novel Non-invasive Technique of Cerebral Compliance and Auto-regulation Assessment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Braincare USA Corp (Industry)
Responsible Party: Principal Investigator, Sergio Brasil, MD, Sergio Brasil, University of Sao Paulo
Other Study IDs: 66721217.0.0000.0068
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Intracranial Hypertension
Keywords: intracranial pressure; transcranial Doppler; jugular compression; cerebral compliance
MeSH Terms: conditions — Intracranial Hypertension | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transcranial Doppler (TCD) ultrasound monitoring — TCD monitoring comatose patients in ICU looking for signs of impaired cerebral compliance
Diagnostic Test: Non invasive intracranial compliance monitoring — A sensor of cardiac beat by beat cranial dilation will be used for monitoring intracranial compliance, in non-invasive fashion.

SUMMARY:
Introduction: Intracranial pressure (ICP) monitoring is essential in several medical situations, however, currently there is an invasive technique, costly, not widely available and sometimes contraindicated. Transcranial Doppler (TCD) pulsatility index (PI) measure can provide indirect information on the cerebrovascular resistance (CVR) augmentation, which is present concomitantly with intracranial hypertension (ICH). The hypothesis that PI measure accurately indicates cerebral compliance impairment (CCI) has been not assessed by large studies currently, and would be of value as a non invasive technique to denote earlier installing of therapeutics to prevent the effects of ICH. Likewise, a novel technique of intracranial compliance assessment by means of an external sensor has been developed, still in need of being prospectively studied.

Objective: The present study aims to assess PI accuracy indicating CCI, and dynamic cerebral auto regulation (dCAR) during internal jugular veins (IJVs) compression observed by both invasive and non-invasive techniques.

Methods: A prospective, observational controlled study, including critical neurological patients with ICP monitoring in normal range (under 20 mmHg). Initially, dCAR is monitored, then, the IJVs are compressed for 60 seconds with ultrasound guidance. We evaluate optic nerve sheath prior to intervention, and dCAR, ICP values, ICP waveforms and PI variation at different times, correlating results.

DETAILED DESCRIPTION:
Introduction

Multimodal monitoring in neurocritical care is essential in current practice. It aims to early Identify treats occurring in the brain of comatose patients and implement targeted therapies to avoid further complications and poorer outcomes.

Some of the methods used for monitoring require invasive procedures, such as the assessment of intracranial pressure (ICP) with intracranial catheter. However, these techniques can raise morbidity, are costly, and are not available or contraindicated1. In addition, the invasive ICP method is not perfectly accurate with cases in which, intracranial hypertension (ICH) may be present despite normal screen ICP values2.

Transcranial Doppler (TCD) is a noninvasive bedside ultrasound technique which could be implemented in the monitoring of raised ICP3-4 and in the identification of impaired intracranial compliance by the compression of the internal jugular veins (IJVs)1. However, such application of the method has not been validate with large prospective studies. Validation of this technique would be of value for screening patients prior to suffer the consequences of ICH.

Recently, a non-invasive cranial strain gauge sensor has been developed, able to provide the curves of cardiac beat by beat cranial dilation. The sensor registers have been demonstrated to be similar to those obtained by the invasive ICP catheters, although large series comparing both techniques are lacking.

Objectives

1) Evaluate the reliability of TCD during the IJVs compression in the assessment of intracranial compliance; 2) evaluate dynamic cerebral auto regulation (dCAR) during IJVs compression. 3) Evaluate the suitability of novel non-invasive intracranial compliance system.

Methods

This is a prospective observational study which will be performed at "Hospital das Clinicas" (São Paulo University School of Medicine). The sample desired is of 50 consecutive subjects, as a pilot study based in recommendations of the literature5. After ethics committee approval, neurological patients of any cause, gender or age, whose underwent ICP monitoring displaying both ICP curves and values will be included. The non-invasive system of intracranial compliance monitoring (Brain4Care Brasil, São Carlos, Brazil) will be used concomitantly. We will exclude patients without insonation window.

The control group will be of healthy subjects, to evaluate PI and cerebral auto-regulation during IJVs compression.

Initially, the study of dynamic cerebral auto regulation through the relationship of spontaneous fluctuations of cerebral blood flow velocity in the middle cerebral arteries (MCAs) and arterial blood pressure, will be done using TCD (DWL Doppler Box 2 MHz, Germany) for five minutes, plus the optic nerve sheath measure (Sonosite Micromaxx 13 MHz, USA), then, ultrasound guided (Sonosite Micromaxx 13 MHz, USA) IJVs compression will be performed for 60 seconds in the included patients, and the following variables will be registered prior and after intervention: blood pressure, mean arterial blood pressure, heart rate, breathing rate, hemoglobin, hematocrit, carbon dioxide pressure (pCO2), oxygen saturation, systolic flow velocity, diastolic flow velocity, mean velocity, pulsatility index, ICP values and changes in the ICP relation P1-P2 (waveform behavior).

One researcher (SB) will perform TCD examinations and obtain patients data, while two blinded researchers (RN and MLO) the offline analysis.

Data will be presented as mean ± standard error of the mean or median and interquartile ranges depending on the nature of the variable. The Chi-square test (χ2) will be used to assess the difference in sex distribution and etiology between groups. To evaluate the homogeneity of the sample we will use the Lèvene test. And, we will use the Kolmogorov-Smirnov test to evaluate the normality of distribution of each variable studied. According to the homogeneity and normality of distribution (Gaussian) of the studied variable will be used the appropriate statistical test (parametric or non-parametric) for each variable. In the homogeneous and Gaussian variables during rest, the analysis of variance (ANOVA) of a factor will be used to test the differences between the groups. In cases of significant F, the Scheffé post-hoc test will be performed for multiple comparisons. In non-homogeneous and / or non-Gaussian variables during rest, the Kruskal-Wallis test will be used, followed by the Dunn's test between the groups. On the other hand, in the homogeneous and Gaussian variables analyzed during the physiological maneuvers, the analysis of variance (ANOVA) of two factors will be used to test the differences between groups. In cases of significant F, the Scheffé post-hoc test will be performed for multiple comparisons. However, in non-homogeneous and / or non-Gaussian variables analyzed during physiological maneuvers, the Wilcoxon (paired data) and Mann-Whitney (unpaired data) tests, when appropriate, will be used. Will be considered as statistically significant to differences with P values <0.05.

ELIGIBILITY:
Inclusion Criteria:

Patients whose underwent ICP monitoring displaying both ICP curves and values.

Exclusion Criteria:

Patients whose display absence of insonation window

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neurological patients (GCS 5 and under) of any cause, gender or age.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Impaired cerebral compliance | 10 minutes
  Performing ICP and TCD monitoring simultaneously during jugular compression, matching waveform behavior through computer software QL Online

SECONDARY OUTCOMES:
Impaired cerebral auto-regulation | 10 minutes
  The same procedure detailed above, matching mean arterial pressure and CBFv in the computer software QL Online
Non-invasive intracranial compliance monitoring | 10 minutes
  The same approaches described above, using the non-invasive Brain4Care system concomitantly.

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dahlqvist MB, Andres RH, Raabe A, Jakob SM, Takala J, Dunser MW. Brain herniation in a patient with apparently normal intracranial pressure: a case report. J Med Case Rep. 2010 Aug 31;4:297. doi: 10.1186/1752-1947-4-297. PMID 20807427
- [Background] Bellner J, Romner B, Reinstrup P, Kristiansson KA, Ryding E, Brandt L. Transcranial Doppler sonography pulsatility index (PI) reflects intracranial pressure (ICP). Surg Neurol. 2004 Jul;62(1):45-51; discussion 51. doi: 10.1016/j.surneu.2003.12.007. PMID 15226070
- [Background] O'Brien NF, Maa T, Reuter-Rice K. Noninvasive screening for intracranial hypertension in children with acute, severe traumatic brain injury. J Neurosurg Pediatr. 2015 Oct;16(4):420-5. doi: 10.3171/2015.3.PEDS14521. Epub 2015 Jul 3. PMID 26140576
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Result] Paschoal FM Jr, Bor-Seng-Shu E, Teixeira MJ. Transcranial Doppler ultrasonography with jugular vein compression can detect impairment of intracranial compliance. Clin Neurol Neurosurg. 2013 Jul;115(7):1196-8. doi: 10.1016/j.clineuro.2012.09.028. Epub 2012 Nov 3. No abstract available. PMID 23128012
- [Derived] Brasil S, Czosnyka M, Paiva WS, Frigieri G. Exploring Cerebrospinal Compensatory Zones Using a Noninvasive Approach. Neurocrit Care. 2025 Dec;43(3):834-841. doi: 10.1007/s12028-025-02320-2. Epub 2025 Jul 14. PMID 40659917
- [Derived] de Moraes FM, Brasil S, Frigieri G, Robba C, Paiva W, Silva GS. ICP wave morphology as a screening test to exclude intracranial hypertension in brain-injured patients: a non-invasive perspective. J Clin Monit Comput. 2024 Aug;38(4):773-782. doi: 10.1007/s10877-023-01120-3. Epub 2024 Feb 14. PMID 38355918
- [Derived] Frigieri G, Robba C, Machado FS, Gomes JA, Brasil S. Application of non-invasive ICP waveform analysis in acute brain injury: Intracranial Compliance Scale. Intensive Care Med Exp. 2023 Jan 27;11(1):5. doi: 10.1186/s40635-023-00492-9. No abstract available. PMID 36703025
- [Derived] Brasil S, Frigieri G, Taccone FS, Robba C, Solla DJF, de Carvalho Nogueira R, Yoshikawa MH, Teixeira MJ, Malbouisson LMS, Paiva WS. Noninvasive intracranial pressure waveforms for estimation of intracranial hypertension and outcome prediction in acute brain-injured patients. J Clin Monit Comput. 2023 Jun;37(3):753-760. doi: 10.1007/s10877-022-00941-y. Epub 2022 Nov 18. PMID 36399214